CLINICAL TRIAL: NCT00623896
Title: Nehb 3-Lead Bipolar Leads for Rapid Diagnosis & Treatment of STEMI
Brief Title: 3 Nehb Precordial Leads Anterior, Dorsalis and Inferior Allow Accurate Diagnostics of Different Heart Conditions
Acronym: Nehb-STEMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Ilya Litovchik, MD, Assaf Harofeh Medical Center Cardiology Institute
Other Study IDs: 174/07
Record Dates: First submitted 2008-02-17; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2007-06

CONDITIONS: Acute Myocardial Infarction With ST Segment Elevation
Keywords: Nehb; ST Elevation Myocardial Infarcton; STEMI; ECG
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The method of ECG recording with the use of three bipolar leads A (anterior), D dorsalis) and J (or I - inferior) was introduced in 1938 by German electrophysiologist W. Nehb. Being positioned on the chest in the immediate proximity to the heart, and being aligned to the anatomic position of the heart, these leads are very sensitive and allow accurate diagnostics of different heart conditions. All the active leads are placed on anterolateral plane of the chest wall requiring little anatomical window making this technique convenient for express diagnostics using compact electrocardiographic devices without any loss of valuable information.

Active electrodes are located on the chest in the following order: 1st- red standard electrode placed in the second intercostal space to the right from sternum corresponding to V1 for standard 12-lead ECG recording, 2nd- green standard lead placed in the position corresponding to V4; 3rd- yellow in the position V7. Then ECG recorded as if in the I standard lead would be defined as Nehb's D, which records the potential on the posterior left ventricle wall; II standard lead would produce Nehb's A which corresponds to the potential on the anterior wall of the left ventricle, and III standard lead would record Nehb's J, which reflects the potential on the diaphragmatic surface of heart.

Been simple and informative, this ECG recording modality may be applicable for usage with compact portable cardiographer devices for express diagnosis in different situations and may allow faster and more adequate outpatient response in the case of emergencies.

Nehb 3 leads ECG can provide the clinician with portable, reliable, comprehensive and constant ECG monitoring and by this facilitate rapid diagnosis and treatment of STEMI.

DETAILED DESCRIPTION:
General Objective: to compare the diagnostic ability of Nehb 3 lead ECG and standard 12 lead ECG in patients presenting to EMS with STEMI.

Inclusion criteria:

Age ≥ 18 years ST elevation in more than 2 contiguous leads (> 1 mV in limb leads & V5-V6; more than 2 mm in V1-V4) Complains of chest, neck, jaw, arm, epigastric or back pain or dyspnea Patients directly transferred to the coronary care unit.

Exclusion criteria:

Unconscious patients Unwillingness to participate in the study Presence of LBBB

Protocol:

100 patients with STEMI will be included. After initial 12 leads ECG made by EMS personnel will show changes consistent with STEMI, a portable Nehb 3 leads (ECG MiniMonitor CG 5000 N) recorder will be connected to the patient. 12 leads ECG recording will be performed according to the EMS and the CCU practices, i.e: before transport, on admission, before and after reperfusion therapy (thrombolysis or PCI), during angina episodes, and every 24 hours since admission. Nehb tracing will be recorded in parallel with standard 12 leads ECG.

ECG findings of standard 12 leads ECG and Nehb 3 leads ECG will be compared for:

Presence of ST elevation (defined as presence of ST segment elevation in 2 or more contiguous leads in 12 leads ECG versus presence of ST segment elevation or depression in 1 or more leads in Nehb ECG).

Area at risk [8] (defined as sum of amplitudes of ST segment elevations of all leads that demonstrate this in 12 leads ECG versus sum of amplitudes of ST segment elevations of all leads in Nehb ECG)

Severity of ischemia [8] (defined as disappearance of S waves in leads with normally negative QRS or J point elevation over more than 50% of R wave height in leads with normally positive QRS in 12 leads versus Nehb ECG)

Time discrimination (defined as presence of ST segment elevation at any time of recording and total amount of such events by 12 leads ECG versus Nehb ECG).

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years
2. ST elevation in more than 2 contiguous leads (> 1 mV in limb leads & V5-V6; more than 2 mm in V1-V4)
3. Complains of chest, neck, jaw, arm, epigastric or back pain or dyspnea
4. Patients directly transferred to the coronary care unit.

Exclusion criteria:

1. Unconscious patients
2. Unwillingness to participate in the study
3. Presence of LBBB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All STEMI Patients admitted to ICCU during the study period with ST elevations presenting on first 12 lead ECG performed on admition.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-05 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Evidence of ST Elevations in Nehb Tracing in all patients with determined STEMI in Standard 12-leads ECG. | On patients' admition to EMS/ICCU

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Litovchik, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center Intensive Coronary Care Unit, Ẕerifin, Israel

REFERENCES:
- [Background] Nehb W. Zur Standardisierung der Brustwandableitungen des Elektrokardiogrammen. Kin. Wochenschz. 17 (1938):1807-1811.// Pollock, P. A comparison of Nehb's bipolar chest leads and the standard 12-lead electrocardiogram in cases of myocardial infarction. American Heart Journal, Research Assistant in Medicine. (1955) 68-71.// De Luca et al: Time Delay to Treatment and Mortality in Primary Angioplasty for Acute Myocardial Infarction: Every Minute of Delay Counts. Circulation 109 (2004): 1224// Atar et al: Electrocardiographic Diagnosis of ST-elevation Myocardial Infarction. Cardiol Clin 24 (2006) 343-365// V. N. Dhruva et al: ST-Segment Analysis Using Wireless Technology in Acute Myocardial Infarction (STAT-MI) Trial J. Am. Coll. Cardiol. 2007;50;509-513//